CLINICAL TRIAL: NCT06577571
Title: A Study of CKM-EMPOWER: Empowering Medical Professionals on CKM With Educational Resources
Brief Title: Testing Educational Videos on Conservative Kidney Management
Acronym: CKM-EMPOWER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment, insufficient funds
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Susan Wong, Associate Professor of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STUDY00020971
Record Dates: First submitted 2024-08-05; First posted 2024-08-29 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Kidney Disease, Chronic
Keywords: Education; Conservative Kidney Management; Provider training
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CKM-EMPOWER (Experimental): Training videos
  Interventions: Other: CKM-EMPOWER
- Usual education (No Intervention): No training videos

INTERVENTIONS:
Other: CKM-EMPOWER — CKM-EMPOWER is a series of 11 just-in-time educational videos on topics related to caring for patients who opt for CKM: CKM overview, dysgeusia, fatigue, restless leg syndrome, uremic pruiritis, cramping, pain, volume overload, electrolyte abnormalities, anticipatory grief, and actively dying patient. Videos are approximately 5-10 minutes in length and intended to provide learners with a brief overiew on the definition of each issue, impact of the issue on a patient, assessment of the issue, and approaches to addressing the issue. Videos conclude with references to additional resources on each topic for more in-depth self-study. CKM-EMPOWER was created by a team comprised of a health educator, the principal investigator (nephrologist), a geriatrician and a physician dually trained in nephrology and palliative care and with feedback from a geriatric pharmacist and members of a national professional interest workgroup in kidney palliative care.
  Arms: CKM-EMPOWER

SUMMARY:
This study aims to test the efficacy of a series of just-in-time educational videos on topics related to CKM (CKM-EMPOWER) in improving nephrology providers ability to provide CKM.

DETAILED DESCRIPTION:
Conservative kidney management (CKM) is an important therapeutic alternative for patients who do not wish to pursue dialysis for their advanced chronic kidney disease (CKD). Despite a growing body of evidence and clinical services to support patients who do not wish to pursue dialysis, nephrologists receive very limited training in CKM. This is a randomized trial of nephrology fellows that utilizes surveys to assess their change in knowledge, confidence and practice of providing CKM with receipt of CKM-EMPOWER. The investigators hypothesize that the CKM-EMPOWER will improve nephrology fellows' knowledge and confidence with delivering key elements of CKM. Investigators will recruit 126 nephrology fellows from US fellowship programs and randomize participants in a 1:1 fashion to either receipt of the CKM-EMPOWER or non-receipt. Participants will complete web-based surveys to assess knowledge and confidence with providing CKM between groups.

ELIGIBILITY:
Inclusion Criteria:

* nephrology fellow enrolled in US nephrology fellowship training program

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-08-27 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in CKM knowledge | 2 weeks
  Number of knowledge questions (total 44) about CKM answered correctly

SECONDARY OUTCOMES:
Confidence with CKM | 2 weeks
  Self-rated confidence scores in practice of 11 different clinical topics related to CKM rated from 1-5, 5 being most confident
Challenges to CKM | 2 weeks
  Self-reported written qualitative description of challenges face with providing CKM
CKM practice change | 2 weeks
  Self-reported written qualitative description of ways in which providers will change the way they provide CKM following receipt of the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-06-07): https://cdn.clinicaltrials.gov/large-docs/71/NCT06577571/Prot_000.pdf